CLINICAL TRIAL: NCT04364555
Title: Efficacy of Topical Treatment With Clobetasol in Symptomatic Oral Lichen Planus. A Multicenter Placebo-controlled Randomized Clinical Trial.
Brief Title: Efficacy of Topical Treatment With Clobetasol in Symptomatic Oral Lichen Planus.
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Malmö University (Other)
Collaborators: Skane University Hospital (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Fredrik Gränse, Dentist, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIKLO-1
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Oral Lichen Planus
Keywords: Oral lichen planus; Treatment; Candida
MeSH Terms: conditions — Lichen Planus, Oral; Torulopsis | interventions — Clobetasol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active/active (Active Comparator): The one bottle for use in the morning has clobetasol-oral gel, and so does the bottle fore use in the evening. The oral cavity will be rinsed with 5ml oral gel during 1 minute. Nystatin will be taken 1ml 4 times daily.
  Interventions: Drug: Clobetasol Propionate
- Placebo/active (Active Comparator): The bottle for use in the morning contains placebo and one for use in the evening contains clobetasol oral gel. The oral cavity will be rinsed with 5ml oral gel during 1 minute. Nystatin will be taken 1ml 4 times daily.
  Interventions: Drug: Placebo/Klobetasol APL oral gel 0.025%
- Placebo/placebo (Placebo Comparator): Both bottles, the one for the morning and the one for use in the evening, contains placebo. The oral cavity will be rinsed with 5ml oral gel during 1 minute. Nystatin will be taken 1ml 4 times daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clobetasol Propionate — Klobetasol APL oral gel 0.025% is a topical steroid for rinsing the oral cavity. Manufactured by APL, Sweden.
  Other Names: Klobetasol APL oral gel 0.025%
  Arms: Active/active
Drug: Placebo/Klobetasol APL oral gel 0.025% — Placebo/active
  Arms: Placebo/active
Drug: Placebo — Placebo/placebo
  Arms: Placebo/placebo

SUMMARY:
The investigators want to study the effect of clobetasol in symptomatic oral lichen planus. The investigators will include 90 patients and randomly allocate them in three groups. The first group will receive active treatment both in the morning an evening. Group two receives placebo in the morning and active treatment in the evening. Group three will get placebo both in the morning and in the evening. All Groups will follow the same protocol with rinsing twice daily with test substance in conjunction with antifungal treatment. The patients will be controlled after two weeks and and again after another two weeks. A biopsy will be performed at inclusion and another biopsy will be taken at the end of the test period. Smears for candida will also be evaluated. The patients will be examined for changes in clinical appearance and will answer questions to note changes in symptoms. Our hypotheses: #Patients receiving clobetasol will have a better resolution af symptoms than those who got placebo. #Patients treated with clobetasol twice daily will have a faster relief of symptoms than patients just treated once daily. #The clinical signs of oral lichen planus will diminish more pronounced in the two groups given active treatment. #A majority of the OLP lesions were infected by candida. #Specific histological changes can be seen in the biopsies taken after clobetasol treatment compared to those taken before treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic oral lichen planus
* Age above 40 years

Exclusion Criteria:

* Lichenoid contact lesions
* Graft versus host disease
* Bacteria related lichenoid reaction
* Intraoral vesiculobullous diseases
* Active antibiotic treatment
* Active treatment with steroids or other immunomodulating substance
* Allergy to Clobetasol
* Severe periodontitis
* Bad oral hygiene
* Biopsy not supporting OLP
* Allergy to nystatin
* Not in menopause
* Previous or actual oral malignancy
* Participation in other medical study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical appearance of the lichen lesion | Four weeks
  Site-, severity- and activity-score according to Escudier et al

SECONDARY OUTCOMES:
Oral health impact profile | Four weeks
  Oral health impact profile (OHIP-14)
Pain score | Four weeks
  VAS scale. A 10 cm scale ranging from no pain what so ever to worst pain imaginable.
Burning sensation score | Four weeks
  VAS scale. A 10 cm scale ranging from no burning sensation what so ever to worst burning sensation imaginable.
Histological appearance | Four weeks
  Amount and degree of lichenoid reaction in biopsy
Candida | baseline (At treatment start)
  Candida hyphae in smear from lichen lesions

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Götrick, Docent, Study Chair — Malmö University
Locations (2):
- Sweden (2):
  - Oral surgery, Universityhospital of Scania, Lund
  - Oral Surgery and oral medicine, Malmö University, Malmo

IPD SHARING:
Plan to Share IPD: No
Still undecided since we dont know what data to share and how, yet.